CLINICAL TRIAL: NCT04803331
Title: Superparamagnetic Iron Oxide-enhanced Magnetic Resonance Imaging for Sentinel Lymph Node Identification in Oral Cancer: a Feasibility Study
Brief Title: SPIO-enhanced MRI in Oral Cancer for Sentinel Lymph Node Identification
Acronym: MAG-NODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAG-NODE study
Record Dates: First submitted 2021-03-04; First posted 2021-03-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Sentinel lymph node identification; Magnetic resonance imaging; Superparamagnetic iron oxide; Oral cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cT1-2N0M0 oral cancer patients (Experimental): Patients undergo routine sentinel lymph node procedure (99mTc injection, planar imaging, SPECT-CT and surgery) for clinical purposes. After 99mTc injections and imaging has been executed peritumoral SPIO injections are performed by a medical doctor. A T2*-weighted iron sensitive MRI scan is made 1 hour later.
  Interventions: Diagnostic Test: SPIO-enhanced MRI

INTERVENTIONS:
Diagnostic Test: SPIO-enhanced MRI — SPIO is peritumorally injected. A T2*-weighted iron sensitive MRI scan is performed 1 hour later to localize and assess the sentinel lymph nodes.

SUMMARY:
To explore the feasibility of sentinel lymph node identification by SPIO injection followed by MRI in head-and-neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >18 years.
* Patients with histopathologically proven cT1-2N0M0 squamous cell carcinoma of the oral cavity.
* Patients planned to undergo routine sentinel node biopsy with 99mTc-radioisotope and SPECT-CT.
* Patient provided written informed consent.

Exclusion Criteria:

* Patients who underwent previous surgery or radiotherapy to the neck.
* Contra-indications to SPIO (Hypersensitivity to iron oxide or dextran compounds, Presence of iron overload disease (hereditary hemochromatosis, hemosiderosis, chronic hemolytic anemia (e.g. thalassemia, sickle cell anemia))
* Contra-indications to MRI: Epilepsy, Claustrophobia, Metallic splinters, Pacemaker, pacemaker wires or implanted defibrillator, Implanted magnets in jaw, Metallic Arterial clips (carotid arteries), Pregnancy, Auditory implant, neurogenic bladder stimulator, insulin pump, neurostimulator, baclofen pump, Metallic tissue expander after mastectomy, Cochlear implant, Metallic braces, Other foreign bodies implanted
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
MR (artefact) finetuning for optimization of SPIO dose and timing of MRI | 2 months
  The first two patients will receive a dose of 0.012 ml SPIO. MR-images will be assessed. If this dose provides satisfactory MR-images (good visualization of lymph nodes without disturbing artefacts), subsequent patients will receive the same dose. If the artefact is too large, the dose will be decreased. If visualization is poor, the dose will be increased. The procedure will be repeated with adjusted doses each time in two patients until satisfactory MR-images are obtained.
  The investigators have established timing of MRI 1 hour after SPIO injection. It is assumed that after this time interval SPIO particles have had sufficient time to migrate to the SNs and to be taken up. However, if this interval appears to be too long because 'too many' SNs are visualized the time interval will be shortened. If this interval appears to be too short since no or too little SNs are visualized because SPIO uptake has not taken place yet, the time interval will be lengthened.

SECONDARY OUTCOMES:
Localization of sentinel lymph nodes detected by conventional 99mTC-nanocollloid injection and SPECT-CT and by SPIO injection and MRI | 1 year
  SPIO-enhanced MR-images and SPECT-CT images are compared to investigate whether SPIO-enhanced MRI detects the same sentinel lymph nodes as SPECT-CT.
Comparison of SPIO distribution within a lymph node on MR-images and histopathological staining. | 1 year
  SNs will be localized on T2* weighted SPIO-enhanced in vivo MR-images by a radiologist. Lymph node status will be assessed based on signal intensity. All surgically removed lymph nodes are embedded in a tissue cassette. Histopathological analysis of these lymph nodes includes multiple sectioning, HE staining, immunohistochemistry and iron staining. The MR-images are compared to the pathology slices to see whether the MR signal intensity pattern matches the benign/malignant structure of the lymph node.

CONTACTS AND LOCATIONS:
Overall Officials: J.H.A.M. Kaanders, MD, PhD, Principal Investigator — Radiation Oncology
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heldens GTN, Driessen DAJJ, Dijkema T, Arens AIJ, Zamecnik P, Pegge SAH, Weijs WLJ, van Engen-van Grunsven ACH, Takes RP, Kaanders JHAM, Scheenen TWJ. SPIO-enhanced MRI for sentinel lymph node mapping in oral cancer: a prospective feasibility study. Eur Radiol Exp. 2025 Nov 15;9(1):113. doi: 10.1186/s41747-025-00636-4. PMID 41241690